CLINICAL TRIAL: NCT04413929
Title: International Observational Non-Interventional Retrospective Program for Studying the Efficiency and Safety of Ergoferon in Patients With Influenza and Acute Respiratory Viral Infection (ARVI).
Brief Title: Study on Safety and Effectiveness of Ergoferon in the Treatment of Flu / ARVI in Outpatients.
Acronym: HERMITAGE
Status: Completed | Type: Observational
Sponsor: Materia Medica Holding (Industry)
Responsible Party: Sponsor
Other Study IDs: HERMITAGE
Record Dates: First submitted 2020-05-25; First posted 2020-06-04 (Actual); Results first posted 2021-04-02 (Actual); Last update posted 2021-04-02 (Actual); Status verified 2020-05

CONDITIONS: Viral Respiratory Infection
MeSH Terms: interventions — ergoferon

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Ergoferon: Oral administration in the therapeutic dosage specified in the instructions for medical use.
  Interventions: Drug: Ergoferon

INTERVENTIONS:
Drug: Ergoferon — Oral administration

SUMMARY:
The observational study to get the additional data of the safety and effectiveness of Ergoferon in the treatment of influenza/ARVI in adult and pediatric outpatients.

DETAILED DESCRIPTION:
This observational study is aimed to provide additional safety and effectiveness data for Ergoferon in the treatment of influenza/ARVI in adult and pediatric outpatients, including cases with delayed treatment initiation of illness, and in allergy patients. Routine clinical practice in the management of outpatients with ARVI is to be studied in Azerbaijan, Armenia, Georgia, Kazakhstan, Kyrgyzstan, Mongolia, Tajikistan and Uzbekistan: the demographic characteristics of patients, duration and time points of treatment with the use of Ergoferon, its safety, and the frequency of additional medication.

Scope of the study: 519 general practitioners; 8411 patients. Physical examinations and tests are performed according to local outpatient clinical practice, and to local and international medical care standards.

Data to be collected and analyzed after the completion of treatment:

* demographics (age, gender, and city/town of residence)
* severity of illness (mild, moderate, or severe)
* comorbidities (chronic ENT conditions, chronic obstructive pulmonary disease (COPD), chronic cardiovascular disease, allergic rhinitis/sinusitis, atopic dermatitis/eczema, asthma, or other)
* the time of resolution of infection symptoms (absence of fever - a body temperature below 37.0°С), systemic symptoms (chills, headaches, myalgias, weakness, and loss of appetite), nasal symptoms (nasal congestion/ discharge), laryngeal symptoms (a sore throat, or other), and other symptoms
* illness time points: onset of illness, first visit to the doctor's office, and start of treatment.
* symptomatic therapy (drug name, date prescribed, and date discontinued)
* therapy for bacterial complications (date the antimicrobial drug is prescribed, drug name, diagnosis, hospitalization or no hospitalization required, date of hospitalization)
* serious adverse events (description of the event, causality (related/ not related to Ergoferon), severity, date of the onset, and actions taken)
* efficacy assessment of the Ergoferon treatment (high efficacy: recovery / satisfactory: improvement/ insufficient: no effect) - observational study model: cohort Cohort study is an observation of outcomes in a group of individuals linked by shared characteristics (an acute respiratory viral infections and use of Ergoferon).

ELIGIBILITY:
Inclusion Criteria:

* Data of children from 6 months to 18 years old and adults over 18 years old.
* Diagnosis: Flu / ARVI.
* Axillary temperature above 37.4 °С.
* At least one systemic and/or catarrhal symptom lasting 12 hours to 3 days by the time the doctor is consulted, for which treatment with Ergoferon is prescribed.
* A specific decision of the doctor to prescribe Ergoferon in strict accordance with the indications, regardless of the factor of including patient data in the program.
* CRF, filled by a doctor on the basis of medical documentation, at the end of patient observation.

Exclusion Criteria:

Not applicable.

Ages: 6 Months to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Children from 6 months to 18 years of age and adults over 18 years of age in any gender and demographic proportion.
Sampling Method: Non-Probability Sample
Enrollment: 8411 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

RESULTS

PARTICIPANT FLOW:
Groups:
- Ergoferon: Oral administration in the therapeutic dosage specified in the instructions for medical use: 8 tablets on the first day of treatment (1 tablet every 30 minutes during the first 2 hours, then 3 more tablet intakes with regular intervals in between);from the second day until recovery take 1 tablet 3 times a day. The duration of the reception was regulated by the physician.
Period: Overall Study
Arm/Group | Ergoferon
Started | 8411
Completed | 8411
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Ergoferon
Number analyzed (Participants) | 8411
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Children (age under 18) and adults presented separately. A number of patients did not reported their age (N=337)
  years
    All included patients: number analyzed (Participants) | 8074
    All included patients | 14.43 (15.44)
    Adults: number analyzed (Participants) | 2069
    Adults | 36.75 (14.1)
    Children: number analyzed (Participants) | 6005
    Children | 6.75 (4.59)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: A number of patients (N=220) did not reported their sex
  Participants
    number analyzed (Participants) | 8191
    Female | 4220
    Male | 3971
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Kazakhstan | 2718
  Uzbekistan | 2142
  Azerbaijan | 1015
  Armenia | 390
  Georgia | 329
  Kyrgyzstan | 807
  Mongolia | 451
  Tajikistan | 559

OUTCOME MEASURES:

1. Primary Outcome: Duration of Influenza/ARVI Symptoms.
Description: The time from the onset of treatment with Ergoferon to the resolution of the symptoms, i.e. a body temperature ≤37.0 °С remaining at this level for 24 h (with no further increases throughout the rest of the observation period) in the absence of catarrhal signs and systemic symptoms. Based on Case Report Form data.
Time Frame: through study completion up to 1 month
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Ergoferon
Number analyzed (Participants) | 8411
days | 4.84 (1.53)

2. Secondary Outcome: Duration of Increased Body Temperature.
Description: A body temperature ≥37.0 °С. Based on Case Report Form data.
Time Frame: through study completion up to 1 month
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Ergoferon
Number analyzed (Participants) | 8411
days | 1.99 (0.87)

3. Secondary Outcome: Duration of Systemic Symptoms.
Description: Symptoms of intoxication (chills, headache, muscle pain, weakness, loss of appetite).
  Based on Case Report Form data.
Time Frame: through study completion up to 1 month
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Ergoferon
Number analyzed (Participants) | 8411
days | 2.33 (1.02)

4. Secondary Outcome: Duration of Nose Symptoms.
Description: Symptoms of the nose (nasal congestion, discharge from the nose), other symptoms. Based on Case Report Form data.
Time Frame: through study completion up to 1 month
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Ergoferon
Number analyzed (Participants) | 8411
days | 2.9 (1.23)

5. Secondary Outcome: Duration of Throat Symptoms.
Description: Symptoms of the throat (sore throat, etc.). Based on Case Report Form data.
Time Frame: through study completion up to 1 month
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Ergoferon
Number analyzed (Participants) | 8411
days | 2.9 (1.3)

6. Secondary Outcome: Percentage of Patients With Complications of Influenza/Acute Viral URI.
Description: Patients who got bacterial complications of influenza/acute viral URI, requiring the antibiotics and/or hospitalization during the observation period.
Time Frame: through study completion up to 1 month
Measure: Count of Participants; unit: Participants
Arm/Group | Ergoferon
Number analyzed (Participants) | 8411
Participants | 1241

ADVERSE EVENTS:
Time Frame: Approximately 6 months
Description: The collection of information was carried out in accordance with the legislation of the participating countries for spontaneous reports of AEs within the framework of the existing practice of ARVI management, monitoring of medical researchers was not carried out due to the non-interventional nature of the study.
Groups:
- Ergoferon: Oral administration in the therapeutic dosage specified in the instructions for medical use.
  Ergoferon: Oral administration in the therapeutic dosage specified in the instructions for medical use.
Arm/Group | Ergoferon
All-Cause Mortality (participants affected / at risk) | 0/8411
Serious Adverse Events (participants affected / at risk) | 0/8411
Other Adverse Events (participants affected / at risk) | 0/8411

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-09-30): https://cdn.clinicaltrials.gov/large-docs/29/NCT04413929/Prot_SAP_000.pdf